CLINICAL TRIAL: NCT04187664
Title: Implementation of the Extended Care in High-Risk Surgical Patient (EXCARE) Pathway in High-risk Non-cardiac Surgical Population: Impact on Morbidity and 30-day Mortality
Brief Title: Extended Care in High-Risk Surgical Patient (EXCARE) Pathway in High-risk Surgical Population
Acronym: EXCARE
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2019-0066
Record Dates: First submitted 2019-12-03; First posted 2019-12-05 (Actual); Last update posted 2020-06-26 (Actual); Status verified 2020-06

CONDITIONS: Postoperative Complications; Patient Care Team
Keywords: failure to rescue; high-risk surgical patient
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Quasi-experimental study, nonrandomized, pre-post intervention study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EXCARE Pathway Group (Experimental): The proposed pathway comprises a range of actions that include individual patient-centered risk assessment by the SAMPE Risk Model (30-day probability of death), specialized care in Post-Anesthetic and Intensive Care Units, and also in the surgical wards performed by the nursing, anesthesia, clinic and surgery teams.
  Interventions: Behavioral: Postoperative Monitoring; Diagnostic Test: High-sensitivity cardiac troponin testing

INTERVENTIONS:
Behavioral: Postoperative Monitoring — Nursing and medical staff will monitor patients vital signs and clinical deterioration triggers twice as often as in previous ward care.
Diagnostic Test: High-sensitivity cardiac troponin testing — High-risk patients will have their high-sensitivity cardiac troponin tested preoperatively and daily for the first 48h postoperatively

SUMMARY:
High risk surgical patients are subject to complications that impact rehabilitation time, overall mortality and costs. This project proposes the creation of a post-surgery care pathway called Extended Care in High-Risk Surgical Patients (EXCARE) in the form of coordinated multiprofessional actions dedicated to high-risk non-cardiac surgical patients with the aim of improving the postoperative outcomes. The proposed pathway comprises a range of actions that include individual patient-centered risk assessment by the Anaesthesia and Perioperative Medicine Service (SAMPE) Risk Model (30-day probability of death), specialized care in Post-Anesthetic and Intensive Care Units (ICU), and also in the surgical wards performed by the nursing, anesthesia, clinic and surgery teams.

This is a quasi-experiment in which the clinical effectiveness of the extended care will be analyzed using a before-and-after comparison, the primary outcome being 30-day surgical mortality and postoperative complications at day 7 defined by PostOperative Morbidity Survey (POMS), a reliable and valid survey of short-term postoperative morbidity in major elective surgery. POMS domains evaluated are: pulmonary, infectious, renal, gastrointestinal, cardiovascular, neurological, haematological and wound complications.

Secondary outcomes include 30-day mortality, hospital length of stay, number of Rapid Response Team calls, unplanned postoperative ICU admission, surgical reintervention, failure to rescue and hospital readmission. High-sensitive cardiac troponin (hs-cTn) levels will be measured before surgery and daily until 48 hours postoperatively to identify patients with myocardial injury (defined as any hs-cTn concentration greater than the 99th-percentile upper reference limit).

DETAILED DESCRIPTION:
Study Strengths and Limitations: This is the first study to evaluate the implementation of surgical patient stratification using the SAMPE Risk Model, pioneering the creation of a multidisciplinary care pathway that involves nursing and medical teams, and can be consolidated as a future standard of assistance. The care bundle, using an objective risk communication tool, is expected to integrate the teams involved in the perioperative care, reducing the fragmentation of care and, consequently, postoperative complications. The study is designed to use historical controls (before and after) and is therefore inherently vulnerable to the biases of this design. It will be conducted in a single teaching hospital and referral centre that provides care to patients from across southern Brazil through the national unified health system centre, which can therefore limit its external validity.

ELIGIBILITY:
Inclusion Criteria:

* Age over 16 years;
* Classified as high-risk by the SAMPE Risk Model (30-day mortality >5%);
* Underwent non-cardiac surgeries at the main operating room unit;
* Referred postoperatively to the postanesthesia care unit or intensive care unit.

Exclusion Criteria:

* Patients undergoing procedures performed outside the operating room unit (outpatient, diagnostic, performed under local anesthesia);
* Patients undergoing cardiac surgery with cardiopulmonary bypass and / or referred to the cardiac ICU postoperatively;
* Patients undergoing organ transplantation;
* Low-risk patients (classified as <5% probability of death within 30 days by the SAMPE Risk Model).

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1720 (Estimated)
Dates: Start 2019-01-30 (Actual); Primary Completion 2021-07-31 (Estimated); Study Completion 2021-07-31 (Estimated)

PRIMARY OUTCOMES:
Mortality | 30 days
  In-hospital mortality within 30 days
Postoperative complications | 7 days
  Postoperative complications within 7-days defined by Post-operative Morbidity Survey (POMS) domains

SECONDARY OUTCOMES:
Length of stay (LOS) | 6 months
  Hospital length of stay (days)
Unplanned intensive care unit (ICU) admission | 30 days
  Admission to ICU due to clinical deterioration within 30 days
Calls to rapid response team (RRT) | 30 days
  Number of calls to the RRT within 30 days
Surgical reintervention | 30 days
  Number of surgical reinterventions within 30 days
Hospital readmission | 30 days
  Hospital readmission within 30 days
Failure to rescue | 30 days
  Death after a treatable complication within 30 days
High-sensitivity cardiac troponin levels | 3 days
  High-sensitivity cardiac troponin (hs-cTn) elevation due to myocardial injury (defined as any hs-cTn concentration greater than the 99th-percentile upper reference limit.) 3 categories:
  * Acute myocardial injury due to myocardial infarction (requires at least 1 of the following: symptoms of myocardial ischemia, new ischemic electrocardiographic changes, new ischemic regional wall-motion abnormalities on cardiac imaging, and/or an acute coronary thrombus on coronary angiography) or nonischemic causes (documented nonischemic etiology);
  * Myocardial Injury After Noncardiac Surgery (MINS): myocardial injury caused by ischemia (that may or may not result in necrosis), has prognostic relevance and occurs during or within 30 days after noncardiac surgery.
  * Chronic myocardial injury: stable but elevated troponin.

CONTACTS AND LOCATIONS:
Overall Officials: Luciana Cadore Stefani, PhD, Study Director — Hospital de Clinicas de Porto Alegre
Locations (1):
- Hospital de Clinicas de Porto Alegre, Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Stefani LC, Gutierrez CS, Castro SMJ, Zimmer RL, Diehl FP, Meyer LE, Caumo W. Derivation and validation of a preoperative risk model for postoperative mortality (SAMPE model): An approach to care stratification. PLoS One. 2017 Oct 30;12(10):e0187122. doi: 10.1371/journal.pone.0187122. eCollection 2017. PMID 29084236
- [Background] Writing Committee for the VISION Study Investigators; Devereaux PJ, Biccard BM, Sigamani A, Xavier D, Chan MTV, Srinathan SK, Walsh M, Abraham V, Pearse R, Wang CY, Sessler DI, Kurz A, Szczeklik W, Berwanger O, Villar JC, Malaga G, Garg AX, Chow CK, Ackland G, Patel A, Borges FK, Belley-Cote EP, Duceppe E, Spence J, Tandon V, Williams C, Sapsford RJ, Polanczyk CA, Tiboni M, Alonso-Coello P, Faruqui A, Heels-Ansdell D, Lamy A, Whitlock R, LeManach Y, Roshanov PS, McGillion M, Kavsak P, McQueen MJ, Thabane L, Rodseth RN, Buse GAL, Bhandari M, Garutti I, Jacka MJ, Schunemann HJ, Cortes OL, Coriat P, Dvirnik N, Botto F, Pettit S, Jaffe AS, Guyatt GH. Association of Postoperative High-Sensitivity Troponin Levels With Myocardial Injury and 30-Day Mortality Among Patients Undergoing Noncardiac Surgery. JAMA. 2017 Apr 25;317(16):1642-1651. doi: 10.1001/jama.2017.4360. PMID 28444280
- [Background] Pearse RM, Moreno RP, Bauer P, Pelosi P, Metnitz P, Spies C, Vallet B, Vincent JL, Hoeft A, Rhodes A; European Surgical Outcomes Study (EuSOS) group for the Trials groups of the European Society of Intensive Care Medicine and the European Society of Anaesthesiology. Mortality after surgery in Europe: a 7 day cohort study. Lancet. 2012 Sep 22;380(9847):1059-65. doi: 10.1016/S0140-6736(12)61148-9. PMID 22998715
- [Background] Ferraris VA, Bolanos M, Martin JT, Mahan A, Saha SP. Identification of patients with postoperative complications who are at risk for failure to rescue. JAMA Surg. 2014 Nov;149(11):1103-8. doi: 10.1001/jamasurg.2014.1338. PMID 25188264
- [Background] Bennett-Guerrero E, Welsby I, Dunn TJ, Young LR, Wahl TA, Diers TL, Phillips-Bute BG, Newman MF, Mythen MG. The use of a postoperative morbidity survey to evaluate patients with prolonged hospitalization after routine, moderate-risk, elective surgery. Anesth Analg. 1999 Aug;89(2):514-9. doi: 10.1097/00000539-199908000-00050. PMID 10439777
- [Derived] Stahlschmidt A, Passos SC, Dornelles DD, Polanczyk C, Gutierrez CS, Minuzzi RR, Castro SMJ, Stefani LC; and the Ex-Care Collaborative. Troponin elevation as a marker of short deterioration and one-year death in a high-risk surgical patient cohort in a low and middle income country setting: a postoperative approach to increase surveillance. Can J Anaesth. 2023 Nov;70(11):1776-1788. doi: 10.1007/s12630-023-02558-4. Epub 2023 Oct 18. PMID 37853279
- [Derived] Stahlschmidt A, Passos SC, Cardoso GR, Schuh GJ, Gutierrez CS, Castro SMJ, Caumo W, Pearse RM; Ex-Care collaborative; Stefani LC. Enhanced peri-operative care to improve outcomes for high-risk surgical patients in Brazil: a single-centre before-and-after cohort study. Anaesthesia. 2022 Apr;77(4):416-427. doi: 10.1111/anae.15671. Epub 2022 Feb 15. PMID 35167136